CLINICAL TRIAL: NCT03291665
Title: Comparing Thickness of the Plantar Fascia in Stretched and Relaxed Positions and the Association With Pressure Pain Threshold in Patients With Plantar Fasciopathy
Brief Title: Thickness of the Plantar Fascia in Stretched and Relaxed Positions in Patients With Plantar Fasciopathy
Status: Completed | Type: Observational
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Henrik Riel, PhD student, Aalborg University
Other Study IDs: 59700
Record Dates: First submitted 2017-09-18; First posted 2017-09-25 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Plantar Fasciopathy
Keywords: Plantar Fasciitis; Plantar heel pain
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will compare the thickness of the plantar fascia in stretched and relaxed positions in patients with plantar fasciopathy using ultrasonography.

DETAILED DESCRIPTION:
The purpose of this observational study is to compare the thickness of the plantar fascia in stretched and relaxed positions of the most symptomatic heel in patients with plantar fasciopathy using ultrasonography.

In addition to this, we will compare measurements of the thickness of the plantar fascia in sagittal versus transversal transducer positions, compare pressure pain thresholds at the most tender spot of the plantar fascia in stretched and relaxed position using pressure algometry and investigate the association between the thickness of the plantar fascia and the pressure pain threshold. All measurements are performed bilaterally starting with the most symptomatic foot.

To compare thickness and pressure pain thresholds in stretched and relaxed positions of the plantar fascia paired-t-tests are used. To compare the most and least symptomatic sides paired-t-tests will be used.

The association between the thickness of the plantar fascia and pressure pain threshold will be investigated using the Pearson's correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

* History of plantar heel pain of at least 3 months
* Clinical presentation of pain and/or tenderness to palpation in the area of the medial tubercle of the calcaneus
* Average intensity of pain in the previous week equal to or greater than 3 on an 11-point visual analog scale (VAS)
* Thickness of symptomatic plantar fascia of 4 mm or greater

Exclusion Criteria:

* Age under 18
* Pregnancy
* History of systemic disease with manifestations similar to those of plantar fasciopathy
* Pain medication in the last 24 hours
* Steroid injection for plantar fasciopathy in the previous 6 months
* Previous heel surgery or fracture of the lower leg or foot

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients from the local community of the municipality of Aalborg, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
Thickness of the plantar fascia in sagittal plane | Immediately after eligibility has been confirmed
  The thickness will be measured in mm in stretched and relaxed positions using ultrasonography with a sagittal transducer position.

SECONDARY OUTCOMES:
Pressure pain threshold | Immediately after eligibility has been confirmed
  Measured in kPa at the most tender spot of the plantar fascia in stretched and relaxed position using pressure algometry. In non-symptomatic feet the antero-medial part of the calcaneus is used as the test site.
Thickness of the plantar fascia in transversal plane | Immediately after eligibility has been confirmed
  The thickness will be measured in mm in stretched and relaxed positions using ultrasonography with a transversal transducer position

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Riel, M.Sc., Study Director — Research Unit for General Practice in Aalborg, Department of Clinical Medicine, Aalborg University
Locations (1):
- Research Unit for General Practice, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ostermann S, Olesen JL, Holden S, Riel H. Stretching and relaxing the plantar fascia may change plantar fascia thickness but not pressure pain thresholds: a cross-sectional study of patients with plantar fasciopathy. BMC Musculoskelet Disord. 2020 Dec 3;21(1):804. doi: 10.1186/s12891-020-03833-x. PMID 33272236